CLINICAL TRIAL: NCT04073238
Title: The Clinical Trial of Myopia Control in Schoolchildren Using the Repeated Low-Level Red-Light Therapy
Brief Title: Efficacy of Repeated Low-Level Red-Light Therapy in Myopia Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: Shenzhen Children's Hospital (Other Government); The Second People's Hospital of Foshan (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019KYPJ093
Record Dates: First submitted 2019-08-18; First posted 2019-08-29 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Myopia; Refractive Errors; Eye Diseases
MeSH Terms: conditions — Myopia; Refractive Errors; Eye Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single vision spectacle lens (No Intervention): Single vision lens with power for correcting distance refraction.
- Repeated low-level red-light therapy (Experimental): Single vision lens & repeated low-level red-light therapy
  Interventions: Device: Low-level Red-light Therapy

INTERVENTIONS:
Device: Low-level Red-light Therapy — In addition to wearing single vision spectacle lens with power for correcting distance refraction, low-level red-light therapy is performed twice per school day at home with an interval of at least 4 hours, each treatment lasting 3 minutes.
  Arms: Repeated low-level red-light therapy

SUMMARY:
The purpose of this study is to determine if repeated low-level red-light therapy can slow myopia progression in Chinese schoolchildren.

DETAILED DESCRIPTION:
Low level light therapy (LLLT) is an innovative and non-invasive therapeutic treatment for a variety of eye diseases. Its potential mechanisms of improving choroidal metabolic rate and circulation may improve scleral hypoxia, thus slowing down the progression of myopia. The investigator's preliminary case-series study suggested that repeated low-level red-light therapy was effective in slowing myopia progression without any clinically observable side effects. Using a randomized clinical trial design, the purpose of this study is to determine if repeated low-level red-light therapy can slow myopia progression in Chinese schoolchildren. Study subjects will be randomly assigned to either the treatment group (receive repeated low-level red-light therapy) or the control group (wearing ordinary single vision lenses). Axial length and cycloplegic refraction will be monitored over one year (1st month, 3rd month, 6th month and 12th month), after which changes in axial length and refractive errors in the two groups will be compared. An interim analysis will be performed at the 3rd month, at which the data will be reported and presented. Appropriate adjustment of the p-value and decision on the continuation of the study will be made.

ELIGIBILITY:
Inclusion Criteria:

1. Age at enrolment: 8-13 years
2. Spherical equivalent refractions (SERs): -1.00 to -5.00 diopters (D)
3. Astigmatism of 2.50 D or less
4. Anisometropia of 1.5 D or less
5. Spectacle corrected monocular logMAR visual acuity (VA): 0 or better
6. Parents' understanding and acceptance of random allocation of grouping

Exclusion Criteria:

1. Strabismus and binocular vision abnormalities in either eye
2. Ocular abnormalities in either eye or other systemic abnormalities
3. Prior treatment of myopia control, e.g. drugs, orthokeratology, progressive addition lenses, bifocal lenses, etc in either eye
4. Other contraindications in either eye

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 264 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Axial length change (mm) | 1 month, 3 months, 6 months and 1 year
  Axial length change (mm) is characterized as the difference between each follow-up visit and baseline values. The IOLMaster is used to measure axial length (mm).

SECONDARY OUTCOMES:
Cycloplegic spherical equivalent change (Diopter) | 1 month, 3 months, 6 months and 1 year
  Cycloplegic spherical equivalent change (Diopter, D) is characterized as the difference between each follow-up visit and baseline values. Cycloplegia is induced with one drop of Alcaine 0.5% followed by two drops of 1% cyclopentolate administered at 0, 5th to each eye. The third drop of cyclopentolate is used if the light reflex exists after 20 minute. The light reflex and pupil dilation is checked after an additional 15 minutes. Dilation and light reflex status is recorded and full cycloplegia is justified if the pupil dilates to 6 millimeters or greater and the light reflex is absent. Refraction is performed with an auto-refractor. The data on spherical and cylindrical power and axis is automatically extracted from the auto-refractor. The spherical equivalent power (D) is calculated as the spherical power (D) plus half of the cylindrical power (D).
Corneal curvature change (mm) | 1 month, 3 months, 6 months and 1 year
  Corneal curvature (mm) is characterized as the difference between each follow-up visit and baseline values. The IOLMaster is used to measure corneal curvature (mm).
Anterior chamber depth change (mm) | 1 month, 3 months, 6 months and 1 year
  Anterior chamber depth (mm) is characterized as the difference between each follow-up visit and baseline values. The IOLMaster is used to measure anterior chamber depth (mm).
White to white change (mm) | 1 month, 3 months, 6 months and 1 year
  White to white (mm) is characterized as the difference between each follow-up visit and baseline values. The IOLMaster is used to measure white to white (mm).
Visual acuity change | 1 month, 3 months, 6 months and 1 year
  Visual acuity change is characterized as the difference between each follow-up visit and baseline values. An ETDRS chart (Precision vision, Villa Park, Illinois, USA) with standard illumination is used to measure distance visual acuity. Visual acuity measurement is performed at a distance of 4 meters. Uncorrected visual acuity is measured for all children.
Incidence of treatment-emergent adverse events | 1 month
  Incidence of treatment-emergent adverse events is the rate of treatment-emergent adverse events over a specified period for subjects in the intervention arm. Subjects are asked to report any treatment-emergent adverse events, including but not limited to glare, flash blindness, and afterimages.
Incidence of treatment-emergent adverse events | 3 months
  Incidence of treatment-emergent adverse events is the rate of treatment-emergent adverse events over a specified period for subjects in the intervention arm. Subjects are asked to report any treatment-emergent adverse events, including but not limited to glare, flash blindness, and afterimages.
Incidence of treatment-emergent adverse events | 6 months
  Incidence of treatment-emergent adverse events is the rate of treatment-emergent adverse events over a specified period for subjects in the intervention arm. Subjects are asked to report any treatment-emergent adverse events, including but not limited to glare, flash blindness, and afterimages.
Incidence of treatment-emergent adverse events | 1 year
  Incidence of treatment-emergent adverse events is the rate of treatment-emergent adverse events over a specified period for subjects in the intervention arm. Subjects are asked to report any treatment-emergent adverse events, including but not limited to glare, flash blindness, and afterimages.

OTHER OUTCOMES:
Axial length change (mm) | 2 years
  Axial length change (mm) is characterized as the difference between 2-year follow-up visit and baseline values. The IOLMaster is used to measure axial length (mm).
Cycloplegic spherical equivalent change (Diopter) | 2 years
  Cycloplegic spherical equivalent change (Diopter, D) is characterized as the difference between 2-year follow-up visit and baseline values. Cycloplegia is induced with one drop of Alcaine 0.5% followed by two drops of 1% cyclopentolate administered at 0, 5th to each eye. The third drop of cyclopentolate is used if the light reflex exists after 20 minute. The light reflex and pupil dilation is checked after an additional 15 minutes. Dilation and light reflex status is recorded and full cycloplegia is justified if the pupil dilates to 6 millimeters or greater and the light reflex is absent. Refraction is performed with an auto-refractor. The data on spherical and cylindrical power and axis is automatically extracted from the auto-refractor. The spherical equivalent power (D) is calculated as the spherical power (D) plus half of the cylindrical power (D).
Visual acuity change | 2 years
  Visual acuity change is characterized as the difference between 2-year follow-up visit and baseline values. An ETDRS chart (Precision vision, Villa Park, Illinois, USA) with standard illumination is used to measure distance visual acuity. Visual acuity measurement is performed at a distance of 4 meters. Uncorrected visual acuity is measured for all children.
Changes in other ocular parameters | 2 years
  The IOLMaster is used to measure ocular parameters (e.g., corneal curvature change). Change of each parameter is characterized as the difference between its 2-year follow-up visit and baseline values.
Incidence of treatment-emergent adverse events | 2 years
  Incidence of treatment-emergent adverse events is the rate of treatment-emergent adverse events over a specified period for subjects in the intervention arm. Subjects are asked to report any treatment-emergent adverse events, including but not limited to glare, flash blindness, and afterimages.

CONTACTS AND LOCATIONS:
Overall Officials: Mingguang He, Professor, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (4):
- China (4):
  - The Second People's Hospital of Foshan, Foshan, Guangdong
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Xiangya Hospital, Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Wang W, Jiang Y, Zhu Z, Zhang S, Xuan M, Tan X, Kong X, Zhong H, Bulloch G, Xiong R, Yuan Y, Chen Y, Zhang J, Zeng J, Morgan IG, He M. Axial Shortening in Myopic Children after Repeated Low-Level Red-Light Therapy: Post Hoc Analysis of a Randomized Trial. Ophthalmol Ther. 2023 Apr;12(2):1223-1237. doi: 10.1007/s40123-023-00671-7. Epub 2023 Feb 15. PMID 36790672
- [Derived] Xiong R, Zhu Z, Jiang Y, Wang W, Zhang J, Chen Y, Bulloch G, Yuan Y, Zhang S, Xuan M, Zeng J, He M. Longitudinal Changes and Predictive Value of Choroidal Thickness for Myopia Control after Repeated Low-Level Red-Light Therapy. Ophthalmology. 2023 Mar;130(3):286-296. doi: 10.1016/j.ophtha.2022.10.002. Epub 2022 Oct 11. PMID 36240954